CLINICAL TRIAL: NCT06677723
Title: Differential Effects of High-frequency Versus Low-frequency Exercise Training in Adolescents With Elevated Depressive Symptoms.
Brief Title: High- vs Low-Frequency Exercise for Depression in Adolescents
Acronym: HFEDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Je Bouge Pour Mon Moral (Other)
Responsible Party: Principal Investigator, Fabien Legrand, Principal Investigator, Je Bouge Pour Mon Moral
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Depression_adolescent_1st_step
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RUN_1*60 (Experimental): exercise training including one weekly running session (60-min long) for 3 weeks
  Interventions: Behavioral: physical activity
- RUN_4*15 (Experimental): exercise training including 4 weekly running sessions (15-min long) for 3 weeks
  Interventions: Behavioral: physical activity
- CONTROL (No Intervention): control group

INTERVENTIONS:
Behavioral: physical activity — moderate-intensity running
  Arms: RUN_1*60; RUN_4*15

SUMMARY:
This research project aims to examine the antidepressant effects of different exercise routines on adolescent depression, which has risen significantly in recent years. Depression, particularly prevalent among adolescents at a global rate of around 12%, is associated with reduced positive emotional responses and difficulties in managing negative emotions. Prior studies indicate that physical activity can boost positive moods, like feelings of excitement and calm, potentially leading to overall mood stabilization with regular exercise. However, results on how exercise influences negative moods remain inconsistent. This study will compare two exercise routines-a single 60-minute weekly session versus four 15-minute weekly sessions of moderate-intensity running-over three weeks to determine which approach has a stronger effect on reducing depressive symptoms in adolescents.

DETAILED DESCRIPTION:
Depression is a mental disorder that affects millions of people globally every year. This mental health issue is particularly prominent in adolescents populations, where depression has been found to increase at a greater rate than in adults over the last decade. In concrete terms, the global current prevalence of depressive disorders (major depressive disorder and dysthymia) is about 7-8% in adults worldwide, whereas it is around 12% among adolescents.

Depression is characterized by a limited capacity to inhibit negative emotions and a dampening of positive affective and emotional reactions.

There is strong evidence that physical activity increases pleasant-activated states like excitement and vigor both immediately following a bout of exercise and more accumulatively, and some studies show that physical activity enhances pleasant-deactivated affective states like calmness or relaxation. Over time, these acute affective responses to physical activity may accumulate to chronically regulate core affect. One logical implication of all this is that shorter but more frequent exercise sessions throughout the week will offer repeated doses of mood improvement, leading to a more stable mood over time, which should predict greater reductions in depressive symptoms.

Previous studies have reported inconsistent and inconclusive findings for the influence of physical activity on unpleasant core affects, and the general pattern in previous research is that physical activity has a more pronounced effect on positive affect than negative affect. Although, recent findings suggest that daily moderate to vigorous physical activity can decrease the level of depressed and angry affects in adolescents.

Therefore, the current randomized controlled study aims to compare the antidepressant effects of a 3-week exercise program with either one weekly 60-minute session or four weekly 15-minute sessions of moderate-intensity running among adolescents (in which findings have been mixed to date).

ELIGIBILITY:
Inclusion Criteria:

* baseline PHQ-9 score > 9 (i.e., "moderate depression")

Exclusion Criteria:

* unability to read and understand French language
* specific medical contraindications for physical activity

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
changes in depressive symptoms | PHQ-9 completed the day before and the day after the 3-week long exercise program
  Depression scores will be obtained using the self-report instrument "Patient Health Questionnaire-9" (PHQ-9). This self-report measure has 9 items that assess depressive symptoms. Items are rated on a 4-point scale ranging from 0 to 3. The final score is obtained by adding the score of each item and can range from 0 to 27 with higher scores indicating greater severity of depressive symptoms. A score of 0-4 indicates no depression, scores 5-9 indicate mild depression, 10-14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20 or above indicates severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- JeBougePourMonMoral, Reims, France

IPD SHARING:
Plan to Share IPD: Yes
anonymized full set of raw data (PHQ-9 scores before and after participation) will be made available
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available on reasonable email request as soon as the study will be published in an academic journal
Access Criteria: Researchers wishing to apply for IPD should outlining the research purpose for which they wish to use the data